CLINICAL TRIAL: NCT00000335
Title: Activity Monitoring Assessment of Opiate Withdrawal
Brief Title: Activity Monitoring Assessment of Opiate Withdrawal - 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NIDA-3-0009-4; Y01-3-0009-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2002-12

CONDITIONS: Opioid-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Morphine

INTERVENTIONS:
Drug: Morphine

SUMMARY:
The purpose of this study is to determine if hyperactivity accompanies abrupt opiate withdrawal in heroin addicts, to determine if computerized solid state activity monitors are capable of quantifying hyperactivity, and to quantify the physical and affective symptoms occurring during abrupt withdrawal in heroin addicts and morphine's capacity to alleviate these symptoms.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1995-09-30 (Actual); Primary Completion 1996-03-20 (Actual); Study Completion 1996-05-20 (Actual)

PRIMARY OUTCOMES:
Depression
Anxiety
Withdrawal severity
Activity
Opiate secondary withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deutsch, M.D., Principal Investigator — Washington D.C. Veterans Affairs Medical Center
Locations (1):
- Washington DC VA, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] 1996 CPDD, NIDA Research Monograph